CLINICAL TRIAL: NCT05326607
Title: Pilot Clinical Investigation of Adaptive Eyeglasses for the Correction of Presbyopia
Brief Title: Pilot Clinical Investigation of Adaptative Eyeglasses for the Correction of Presbyopia
Acronym: eve-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laclaree (Industry)
Collaborators: Iris Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A00521-40
Record Dates: First submitted 2022-03-01; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Arm (Other)
  Interventions: Device: Prototype of adaptive eyeglasses; Device: Comparator
- Second Arm (Other)
  Interventions: Device: Prototype of adaptive eyeglasses; Device: Comparator

INTERVENTIONS:
Device: Prototype of adaptive eyeglasses — The tested investigational medical device is a prototype of semi-integrated eyeglasses.
Device: Comparator — The comparator is either a pair of progressive lenses that provide clear vision at both distance and near vision, either, for wearers who have rejected progressive glasses, an alternative solution providing clear vision at both distance and near vision which can consist of bifocal glasses, multifocal or monovision lenses, multiple pairs of glasses or one pair for cases of emmetropia.

SUMMARY:
This study is a pilot clinical investigation of adaptive eyeglasses for the correction of presbyopia. The goal of this clinical investigation is to assess IMD safety and to obtain patient feedback on the usefulness of the Laclarée eyeglasses, through subjective clinical measures and qualitative evaluations. This is an exploratory investigation.

DETAILED DESCRIPTION:
Presbyopia is a visual impairment caused by the normal aging of the eye lens and resulting in progressive loss of accommodation. As a consequence, from the onset of presbyopia occurring around 40-45 years old, the eye has growing trouble focusing at near and intermediate distances. Millions of presbyopes encounter difficulties with current corrective solutions, leading to vision and postural discomfort. Laclarée's adaptive eyeglasses are providing an alternative solution, closer to the native crystalline accommodation. Besides an enhanced field-of-view, these eyeglasses offer a disruptive ergonomics where the glasses automatically adjust to the wearer's need to provide clear vision at all distances and can be electronically recalibrated to adjust the delivered addition throughout presbyopia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient >18 years of age, male or female who has given explicit informed consent (dated and signed)
2. Diagnosed with presbyopia
3. A wearer whose current corrective solution is a pair of progressive lenses that provide clear vision at both distance and near vision (worn at least 5 times per week for 4 hours per day), or, a wearer who has rejected progressive glasses that provide clear vision at both distance and near vision and who uses another corrective solution that provides clear vision at both distance and near vision (bifocal glasses, multifocal or monovision lenses, multiple pairs of glasses or one pair for cases of emmetropia)
4. Patient with a distance visual acuity of 10/10 at least with current corrective solution
5. Patient with a visual acuity of P2 at least in near vision with current corrective solution
6. Patient with at least 10/10 distance vision once corrected with contact lenses for the test
7. Inter-pupillary distance in distance vision between 55 and 71mm
8. Distance from temple-to-temple not exceeding 161mm
9. Addition greater than or equal to 1.75D: Add≥1.75D
10. Sphere strictly between -6D and +4D: -6D<S<+4D
11. Cylinder below 1.75D:C<1.75D
12. Patient uses a computer (at least 3 times a week in private and/or work settings).
13. Affiliation to a social security scheme
14. French-speaking (fluent).
15. Patient willing to participate in the study.

Exclusion Criteria:

1. Patient under tutorship or guardianship.
2. Patient unable to understand the study procedures and therefore to provide free and informed consent
3. Patient with reading difficulties
4. Patient with multifocal implants
5. Patient who has undergone multifocal surgery
6. Patient with prism correction
7. Patient with a current or past eye condition that may adversely affect vision
8. Patient being treated or having undergone surgery likely to adversely affect vision
9. Patient with mobility problems that would prevent tests and workshops from being carried out
10. Patient intolerant to wearing contact lenses for a few hours (only for presbyopes with ametropia)
11. Patient who is pregnant or breastfeeding
12. Patient already included once in the study
13. Patient placed in an institution based on a judicial or regulatory ruling, held in psychiatric department, in state-run prison, or employed by the study research sites or by the sponsor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
IMD safety evaluation | 2 hours
  To evaluate the IMD safety : Collection of adverse events.

SECONDARY OUTCOMES:
Exploratory evaluation of the IMD - controlled tests assessing visual acuity and performance on visual tasks | 2 hours
  To make an exploratory evaluation of the IMD performance on patient vision quality, when compared to that obtained with the patient usual personal eyewear (comparator) : Subjective measures on controlled tests assessing visual acuity and performance on visual tasks.
Exploratory evaluation of the IMD - a questionnaire assessing vision quality | 2 hours
  To make an exploratory evaluation of the IMD performance on patient vision quality, when compared to that obtained with the patient usual personal eyewear (comparator) : Subjective measures on questionnaires.
Exploratory evaluation of the IMD - patient qualitative feedback | 2 hours
  To make an exploratory evaluation of the IMD performance on patient vision quality, when compared to that obtained with the patient usual personal eyewear (comparator) : Collection of patient feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BERGE, PhD, Study Chair — SPONSOR: LACLAREE; Jessica JAROSZ, PhD, Study Director — SPONSOR: LACLAREE; Philippe GAIN, Prof., Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne Hôpital Nord, Service d'Ophtalmologie 25, boulevard Pasteur, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No
Not planned

REFERENCES:
- See also: Jessica Jarosz, Norbert Molliex, Guilhem Chenon, and Bruno Berge, "Adaptive eyeglasses for presbyopia correction: an original variable-focus technology," Opt. Express 27, 10533-10552 (2019) — https://opg.optica.org/oe/fulltext.cfm?uri=oe-27-8-10533&id=408132
- See also: Jessica Jarosz, Norbert Molliex, Quentin Lavigne, and Bruno Berge "An original low-power opto-fluidic engine for presbyopia-correcting adaptive eyeglasses", Proc. SPIE 10858, Ophthalmic Technologies XXIX, 1085824 (28 February 2019) — https://doi.org/10.1117/12.2507816